CLINICAL TRIAL: NCT04855643
Title: Home-based Transcranial Direct Current Stimulation (tDCS) for Apathy in Alzheimer's Disease and Related Dementias (ADRD)
Brief Title: Home-based tDCS for Apathy in Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved to a new institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Alzheimer's Research and Care Consortium (Other)
Responsible Party: Principal Investigator, Antonio L. Teixeira, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-21-0089
Record Dates: First submitted 2021-04-15; First posted 2021-04-22 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease and Related Dementias
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: home-based active tDCS
- Control Group (Sham Comparator)
  Interventions: Device: home-based sham tDCS

INTERVENTIONS:
Device: home-based active tDCS — Anode and cathode electrodes will be placed over the left and right dorsolateral prefrontal cortexes, respectively, with the use of the Omni-Lateral-Electrode system. Caregivers will set up and administer tDCS for participants with ADRD at home. tDCS will be applied for 30 min at an intensity of 2mA, with 30 s ramping up and down. All sessions will be remotely supervised by trained research staff.
  Arms: Treatment
Device: home-based sham tDCS — For sham stimulation, electric current will be applied only in the first 30s tDCS. All sessions will be remotely supervised by trained research staff.
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess feasibility, acceptability, and safety of providing tDCS to Alzheimer's disease and related dementias (ADRD) patients with apathy and to assess the efficacy of tDCS for ADRD-related symptoms, with a primary focus on apathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible or probable ADRD according to the National Institute of Aging - Alzheimer's Association diagnostic criteria
* Mild or moderate dementia, as defined by a MMSE score between 14 and 26
* Clinically meaningful apathy for at least four weeks, clinically diagnosed according to 2018 Apathy Diagnostic Criteria or defined as Neuropsychiatric Inventory (NPI-Q) apathy score equal or above 4 (i.e., severity of 'moderate' or greater and caregiver distress 'mild' or greater).
* Stable doses of cholinesterase inhibitors, memantine and other psychotropic medications for at least three months.

Exclusion Criteria:

* Unstable medical conditions
* History of epilepsy
* Metallic objects in the brain
* Diagnosis of major depression and/or a score higher than 18 on the Cornell Scale for Depression in Dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio L Teixeira Jr, MD.PhD,MSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira AL, Martins LB, Cordeiro TME, Jose L, Suchting R, Holmes HM, Acierno R, Ahn H. Home-based tDCS for apathy in Alzheimer's disease: a protocol for a randomized double-blinded controlled pilot study. Pilot Feasibility Stud. 2023 May 5;9(1):74. doi: 10.1186/s40814-023-01310-5. PMID 37147739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control Group
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control Group | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 79 (0) | 82 (5) | 81 (4.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3
Comorbidities [Count of Participants; unit: Participants]
  Dyslipidemia | 1 | 2 | 3
  Hypertension | 1 | 2 | 3
  Glaucoma | 0 | 1 | 1
  Osteoarthritis | 1 | 2 | 3
Medications in use [Count of Participants; unit: Participants]
  Aspirin | 0 | 1 | 1
  Atorvastatin | 1 | 1 | 2
  Tamsulosin | 0 | 1 | 1
  Citalopram | 0 | 1 | 1
  Hydrochlorothiazide | 0 | 1 | 1
  Vitamin B12 | 0 | 1 | 1
  Vitamin D | 0 | 1 | 1
  Donapezil | 1 | 1 | 2
  Memantine | 1 | 1 | 2
  Pregabalin | 0 | 1 | 1
  Sertraline | 0 | 1 | 1
  Amlodipine | 1 | 1 | 2
  Rosuvastatin | 0 | 1 | 1
  Cilostasol | 1 | 0 | 1
  Duloxetine | 1 | 0 | 1
  Carvedilol | 1 | 0 | 1
  Clopidogrel | 1 | 0 | 1
  Eliquis | 1 | 0 | 1
Time Since Diagnosis [Mean (Standard Deviation); unit: years] | 3 (0) | 3.5 (1.5) | 3.33 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Included and Who Successfully Completed the Protocol
Description: The feasibility will be assessed based on the recruitment rate (per month), randomization success, blind success, retention, and attrition rates.
Time Frame: through study completion (about 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

2. Primary Outcome: How Satisfied the Participant Was With the Treatment as Measured by the tDCS Experience Questionnaire
Description: Acceptability will be measured using a Likert scale composed by 10 questions, each one ranging from 0 (strongly disagree) to 10 (strongly agree).
  The 10 prompts are as followed:
  1. It was easy to prepare the device and accessories
  2. The device was unnecessarily complex
  3. The device was easy to use
  4. I felt the video conferences with a technical person were helpful
  5. I would imagine that most people would learn to use this device quickly
  6. The device was cumbersome to use
  7. I felt confident using the device
  8. I needed to learn a lot of things before I could get going with this device
  9. The effectiveness of the treatment increased over the course of treatment
  10. Overall, I felt that transcranial electrical stimulation treatment benefited me
Time Frame: Baseline
Population: Data were not collected for this outcome measure.
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: How Satisfied the Participant Was With the Treatment as Measured by the tDCS Experience Questionnaire
Description: as for outcome 2
Time Frame: 2 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  It was easy to prepare the device and accessories | 2 (0) | 10 (0)
  The device was unnecessarily complex | 2 (0) | 0 (0)
  The device was easy to use | 2 (0) | 10 (0)
  I felt the video conferences with a technical person were helpful | 8 (0) | 10 (0)
  I would imagine that most people would learn to use this device quickly | 8 (0) | 10 (0)
  The device was cumbersome to use | 1 (0) | 0 (0)
  I felt confident using the device | 8 (0) | 10 (0)
  I needed to learn a lot of things before I could get going with this device | 5 (0) | 0 (0)
  The effectiveness of the treatment increased over the course of treatment | 2 (0) | 5 (7.07)
  Overall, I felt that transcranial electrical stimulation treatment benefited me | 1 (0) | 5.5 (6.36)

4. Primary Outcome: How Satisfied the Participant Was With the Treatment as Measured by the tDCS Experience Questionnaire
Description: as for outcome 2
Time Frame: 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  It was easy to prepare the device and accessories | 10 (0) | 10 (0)
  The device was unnecessarily complex | 0 (0) | 0 (0)
  The device was easy to use | 9 (0) | 10 (0)
  I felt the video conferences with a technical person were helpful | 8 (0) | 10 (0)
  I would imagine that most people would learn to use this device quickly | 8 (0) | 10 (0)
  The device was cumbersome to use | 9 (0) | 0 (0)
  I felt confident using the device | 10 (0) | 10 (0)
  I needed to learn a lot of things before I could get going with this device | 1 (0) | 0 (0)
  The effectiveness of the treatment increased over the course of treatment | 0 (0) | 7 (4.24)
  Overall, I felt that transcranial electrical stimulation treatment benefited me | 0 (0) | 7 (4.24)

5. Primary Outcome: How Satisfied the Participant Was With the Treatment as Measured by the tDCS Experience Questionnaire
Description: as for outcome 2
Time Frame: 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  It was easy to prepare the device and accessories | 9 (0) | 10 (0)
  The device was unnecessarily complex | 0 (0) | 0 (0)
  The device was easy to use | 9 (0) | 10 (0)
  I felt the video conferences with a technical person were helpful | 10 (0) | 10 (0)
  I would imagine that most people would learn to use this device quickly | 8 (0) | 10 (0)
  The device was cumbersome to use | 7 (0) | 0 (0)
  I felt confident using the device | 10 (0) | 10 (0)
  I needed to learn a lot of things before I could get going with this device | 9 (0) | 0 (0)
  The effectiveness of the treatment increased over the course of treatment | 0 (0) | 1.5 (2.12)
  Overall, I felt that transcranial electrical stimulation treatment benefited me | 0 (0) | 1.5 (2.12)

6. Primary Outcome: How Satisfied the Participant Was With the Treatment as Measured by the tDCS Experience Questionnaire
Description: as for outcome 2
Time Frame: 6 weeks post-treatment (12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  It was easy to prepare the device and accessories | 10 (0) | 10 (0)
  The device was unnecessarily complex | 0 (0) | 0 (0)
  The device was easy to use | 10 (0) | 10 (0)
  I felt the video conferences with a technical person were helpful | 2 (0) | 10 (0)
  I would imagine that most people would learn to use this device quickly | 3 (0) | 10 (0)
  The device was cumbersome to use | 1 (0) | 0 (0)
  I felt confident using the device | 10 (0) | 10 (0)
  I needed to learn a lot of things before I could get going with this device | 1 (0) | 0 (0)
  The effectiveness of the treatment increased over the course of treatment | 10 (0) | 5 (0)
  Overall, I felt that transcranial electrical stimulation treatment benefited me | 0 (0) | 5 (0)

7. Primary Outcome: Safety of Home-based tDCS Treatment as Assessed by Side Effects
Description: Safety will be assessed with a questionnaire about side effects that include itching, burning, headache, fatigue, and dizziness.
Time Frame: From baseline to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
Participants
  Tingling at site of contact with electrodes | 1 | 0
  Burning sensation at site of contact with electrodes | 1 | 0
  Fatigue | 0 | 1
  Difficulty concentrating | 0 | 1
  Mood change | 0 | 1
  Itching at site of contact with electrodes | 0 | 1

8. Secondary Outcome: Apathy as Assessed by the Brief Dimensional Apathy Scale (b-DAS)
Description: This scale consists of 9 questions each one scored from 0 (almost always) to 3 (hardly ever). Total scores are reported by summing all of the item's scores, with a minimum of 0 and a maximum of 27. A high score indicates a worse outcome.
Time Frame: Baseline, treatment week 2 (2 weeks from baseline), treatment week 4 (4 weeks from baseline), treatment week 6 (6 weeks from baseline), and 6 weeks post-treatment (12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  Baseline | 18 (0) | 21 (0)
  Treatment Week 2 (2 weeks from baseline) | 21 (0) | 17.5 (1.5)
  Treatment Week 4 (4 weeks from baseline) | 23 (0) | 13 (5)
  Treatment Week 6 (6 weeks from baseline) | 21 (0) | 17 (2)
  6 weeks post-treatment (12 weeks from baseline) | 24 (0) | 15.5 (5.5)

9. Secondary Outcome: Dementia-related Behavioral Symptoms as Assessed by the Neuropsychiatric Inventory (NPI-Q) Scale (Severity Score)
Description: NPI-Q evaluates 12 discrete neuropsychiatric symptoms considering their severity and the related caregiver distress. The severity score ranges from 0 to 36. A high score indicates a worse outcome.
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  Baseline | 9 (0) | 12.5 (7.5)
  treatment week 2 (2 weeks from baseline) | 5 (0) | 14 (12)
  treatment week 4 (4 weeks from baseline) | 6 (0) | 9.5 (6.5)
  treatment week 6 (6 weeks from baseline) | 10 (0) | 10 (6)
  6 weeks post-treatment (12 weeks from baseline) | 10 (0) | 8.5 (8.5)

10. Secondary Outcome: Dementia-related Behavioral Symptoms as Assessed by the Neuropsychiatric Inventory (NPI-Q) Scale (Caregiver Distress Score)
Description: NPI-Q evaluates 12 discrete neuropsychiatric symptoms considering their severity and the related caregiver distress.The caregiver distress score ranges from 0 to 60. A high score indicates a worse outcome.
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  Baseline | 3 (0) | 13 (6)
  Treatment Week 2 (2 weeks from baseline) | 5 (0) | 11.5 (9.5)
  Treatment Week 4 (4 weeks from baseline) | 5 (0) | 6 (3)
  Treatment Week 6 (6 weeks from baseline) | 6 (0) | 7 (5)
  6 weeks Post-Treatment (12 weeks from baseline) | 6 (0) | 10.5 (10.5)

11. Secondary Outcome: Depressive Symptoms as Assessed by the Cornell Scale for Depression in Dementia
Description: This scale assess depressive symptoms and consists of 19 questions. Each question is scored on a 2-point severity scale: 0 = absent; 1 = mild or intermittent; 2 = severe. Total score range is 0 to 38, with a higher score indicating a worse outcome.
Time Frame: Baseline, treatment week 6 (6 weeks from baseline), and 6 weeks post-treatment (12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  Baseline | 13 (0) | 12 (3)
  treatment week 6 (6 weeks from baseline) | 9 (0) | 8.5 (3.5)
  6 weeks post-treatment (12 weeks from baseline) | 9 (0) | 9 (3)

12. Secondary Outcome: Cognition as Evaluated by the Mini-Mental State Examination (MMSE)
Description: The Mini-Mental State Examination (MMSE) includes memory, language, praxis and orientation tasks, yielding a global cognition score ranging from 0 to 30, with a higher score indicating better performance.
Time Frame: Baseline, treatment week 6 (6 weeks from baseline), and 6 weeks post-treatment(12 weeks from baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  Baseline | 26 (0) | 23.5 (2.5)
  Treatment Week 6 (6 weeks from baseline) | 23 (0) | 25 (1)
  Treatment Week 12 (12 weeks from baseline) | 28 (0) | 24 (4)

13. Secondary Outcome: Apathy as Measured by the Apathy Evaluation Scale (AES)
Description: The Apathy Evaluation Scale (AES) consists of 18 items phrased as questions that are to be answered by the caregiver on a four-point Likert scale (1-4), with a higher score indicating greater severity of apathy. The score ranges from a minimum of 18 to a maximum of 72
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 1 | 2
score on a scale
  Baseline | 32 (0) | 41 (4)
  Treatment Week 2 (2 weeks from baseline) | 38 (0) | 42 (4)
  Treatment Week 4 (4 weeks from baseline) | 43 (0) | 45 (3)
  Treatment Week 6 (6 weeks from baseline) | 41 (0) | 46 (2)
  6 Weeks Post-Treatment (12 weeks from baseline) | 40 (0) | 47 (8)

ADVERSE EVENTS:
Time Frame: 6 weeks post treatment (12 weeks from baseline)
Arm/Group | Treatment | Control Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=1) | Control Group (N=2)
Tingling at site of contact with electrodes (General disorders) | 1 | 0
Burning sensation at site of contact with electrodes (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Difficulty concentrating (General disorders) | 0 | 1
Mood Change (General disorders) | 0 | 1
Itching at site of contact with electrodes (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Did not meet enrollment target, resulting in small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT04855643/Prot_SAP_000.pdf